CLINICAL TRIAL: NCT06541730
Title: A Phase Ic Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of DA-302168S Tablets in Overweight/Obese Subjects After Multiple Oral Administration
Brief Title: A Study Evulating DA-302168S Tablets in Overweight/Obese Subjects
Acronym: DA168
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chendu DIAO Pharmaceutical Group CO., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-CP-DA168-05
Record Dates: First submitted 2024-08-01; First posted 2024-08-07 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DA-302168S (Experimental)
  Interventions: Drug: DA-302168S
- Placebo of DA-302168S (Placebo Comparator)
  Interventions: Drug: Placebo of DA-302168S

INTERVENTIONS:
Drug: DA-302168S — Titration was used in this study, and the initial plan was to dose titration in cohort 1 (15 mg dose group). The titration regimen and titration dose for subsequent cohorts will be determined based on the results of cohort 1, including the starting dose of titration, frequency of administration, and titration amplitude.
  Arms: DA-302168S
Drug: Placebo of DA-302168S — Titration was used in this study, and the initial plan was to dose titration in cohort 1 (15 mg dose group). The titration regimen and titration dose for subsequent cohorts will be determined based on the results of cohort 1, including the starting dose of titration, frequency of administration, and titration amplitude.
  Arms: Placebo of DA-302168S

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of continuous oral administration of DA-302168S tablets for 28 days in overweight/obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~60 years old, male and female.
* Weight: male ≥50 kg, female ≥45 kg, body mass index (BMI) in the range of 24.0 to 35.0 kg/m2.
* Stable weight in the 3 months prior to screening (self-reported weight change less than 5%).
* Subject and his or her spouse or partner did not plan to become pregnant or plan to donate sperm or ovums from 14 days prior to screening to 3 months after the last dose, and agreed to use at least one acceptable method of effective contraception.
* Written informed consent prior to any study specific procedures.

Exclusion Criteria:

* Subjects with secondary obesity, such as obesity caused by metabolic diseases (such as Cushing's syndrome, decreased thyroid function, etc.) or drug-induced obesity (such as glucocorticoids, tricyclic antidepressants, atypical antipsychotics, etc.)
* Subjects with clinically significant cardiovascular and cerebrovascular diseases, including a history of angina pectoris, myocardial infarction, stroke or severe peripheral arterial circulation disorder, or transient ischemic attack within 1 year before signing the ICF; There are risk factors for tip torsion ventricular tachycardia. The presence of untreated severe arrhythmias, such as sick sinus syndrome, second or third degree atrioventricular block; New York Heart Association Heart Function Class II-IV heart failure.
* Previous history or family history of medullary thyroid carcinoma, thyroid C-cell hyperplasia, or multiple endocrine adenomatosis type 2;
* Subjects with acute pancreatitis or acute cholecystitis within 3 months before signing the ICF, or with chronic pancreatitis in the past, a history of symptomatic gallbladder (such as multiple gallstones, etc.), or a history of pancreatic injury and other high-risk factors that may lead to pancreatitis;
* Had any malignancy within 5 years prior to signing the ICF (except cured basal cell carcinoma of the skin or carcinoma in situ of the cervix);
* The presence of concomitant diseases, including but not limited to diseases of the respiratory system, digestive system, nervous system, genitourinary system, blood system, endocrine system, etc. that are determined by the investigator to affect the safety of the subject or the findings of the study;
* Those who had previously undergone weight loss surgery (excluding acupuncture for weight loss, liposuction and abdominal fat removal 1 year before screening) or planned to undergo surgery for obesity during the study period, such as gastric bypass or gastric banding;
* Subjects who have experienced severe hypoglycemia or recurrent symptomatic hypoglycemia (≥2 times within half a year) in the past;
* Subjects who have a history of specific allergies (asthma, urticaria, eczema, etc.) or allergies, or are allergic to any component of the investigatory drug or preparation, or are allergic to other GLP-1RA drugs or drugs that have a mechanism of activating GLP-1 receptor;
* HbA1c≥6.5%, or fasting blood glucose ≥7.0 mmol/L or ≤3.9 mmol/L at screening period, or previously diagnosed with type 1 diabetes, type 2 diabetes, or other specific type of diabetes;
* Subjects with a history of thyroid dysfunction who still need drug therapy at screening, or abnormal thyroid function results at screening that are clinically significant;
* A history of moderate to severe depression, anxiety disorder, or a history of serious mental illness, such as schizophrenia or bipolar disorder; Or previous suicidal tendencies or behaviors;
* A history of dysphagia or any gastrointestinal disorder that affects drug absorption (as determined by the investigator);
* Subjects who cannot tolerate venipunction, have a history of needle fainting and blood fainting;
* Lactose intolerant;
* Those who test positive for drug abuse or have a history of drug abuse in the past five years or have used drugs in the three months prior to screening;
* Subjects who had received a glucose-lowering drug such as GLP-1 receptor agonist, dipeptidyl peptidase-4 (DPP-4) inhibitor, sodium-glucose cotransporter-2 (SGLT-2) inhibitor, insulin, metformin, insulin secretagotropin, or thiazolidinedione (TZD) within 3 months prior to screening;
* Use of drugs that have an impact on body weight in the 3 months prior to screening, including any approved or unapproved weight loss drugs, such as orlistat, lorcasserin, phentermine/topiramate, naltrexone/bupropion, etc.) or Chinese herbs, health products, meal replacements, etc., that affect body weight; Systemic steroid hormone use (intravenous, oral or intra-articular administration), tricyclic antidepressants, psychiatric medications or sedatives (such as imipramine, amitriptyline, mirtazapine, paroxetine, phenethazine, chlorpromazine, thiridazine, clozapine, olanzapine, valproic acid, valproic acid derivatives, lithium salts); Note: Except cumulative or continuous use of systemic sex hormones for less than 14 days;
* Those who have participated in other drug clinical trials and received any drug in clinical trials within 3 months prior to screening;
* Subjects who have donated blood or lost blood ≥400 mL, received blood transfusion or used blood products in the 3 months prior to screening;
* Smokers or smokers who smoked an average of ≥5 cigarettes per day in the 3 months prior to screening, or who could not stop using any tobacco products during the study;
* Alcoholics or regular drinkers in the three months prior to screening, i.e. those who consume more than 14 standard units of alcohol per week (1 unit of alcohol =360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine) or who test positive for blood alcohol at baseline, or who cannot stop using any alcohol-containing products during the test period;
* Untreated or poorly controlled hypertension (defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg) at the screening period
* Mean corrected QT interval (corrected by Fridericia's formula) of the three supine 12-lead ECG measurements was >450 msec;
* Periodclinical laboratory examination (local laboratory) results showed any of the following abnormal subjects (re-confirmed once within 1 week if necessary) : alanine aminotransferase (ALT) ≥2.0× upper limit of normal (ULN); Aspartate aminotransferase (AST) ≥2.0×ULN; Blood total bilirubin (TBIL) ≥1.5×ULN; Amylase or lipase >1.5×ULN; Calcitonin ≥50 ng/L; Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 [CKD-EPI formula, see Appendix 4]; Triglyceride (TG) > 500 mg/dl (5.65 mmol/L);
* Subjects tested positive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCVAb), human immunodeficiency virus antibody (HIVAb), or Treponema pallidum antibody (TP-Ab);
* Female subjects who are pregnant or breastfeeding, or who test positive for pregnancy;
* Those who consumed an average of excessive amounts of tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup =250 mL) per day during the 3 months prior to screening, or had consumed tea, coffee and/or caffeinated beverages within 48 hours prior to initial dosing, or could not stop drinking during the study;
* Subjects who have been chronically consuming drinks or foods rich in xanthine or grapefruit, or who have taken any products rich in xanthine or grapefruit within 48 hours before the first dose;
* Any other factors that might affect the evaluation of the relevant indicators for this study identified by the investigator that were not suitable for participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Through study completion, an average of 49 days.
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Cmax | Day 7 to day 8, day 14 to day 15, day 21 to day 22, day 28.
  Plasma samples were collected at different points for pharmacokinetic analysis.
Tmax | Day 7 to day 8, day 14 to day 15, day 21 to day 22, day 28.
  Plasma samples were collected at different points for pharmacokinetic analysis.
AUC0-t | Day 7 to day 8, day 14 to day 15, day 21 to day 22, day 28.
  Plasma samples were collected at different points for pharmacokinetic analysis.
Cmin | Day 7 to day 8, day 14 to day 15, day 21 to day 22, day 28.
  Plasma samples were collected at different points for pharmacokinetic analysis.
PTR | Day 7 to day 8, day 14 to day 15, day 21 to day 22, day 28.
  Plasma samples were collected at different points for pharmacokinetic analysis.
Swing | Day 7 to day 8, day 14 to day 15, day 21 to day 22, day 28.
  Plasma samples were collected at different points for pharmacokinetic analysis.
Body Weight | Day 1, 8, 15, 22, 29.
  Percentage change in body weight from baseline.
Changes in glycosylated hemoglobin (HbA1c) relative to baseline after 28 days of administration. | Day 1, 29.
  Blood samples will be assessed for HbA1c (glycated hemoglobin)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hu, Doctor, Principal Investigator — The Second Hospital of Anhui Medical University; Yi Jun Du, Doctor, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No